CLINICAL TRIAL: NCT05155631
Title: Sex Related Differences in the Effect of Cognitive Behavioral Therapy (CBT) on Emotional Arousal and Salience Circuits and the Role of the Gut Microbiome
Brief Title: Sex Differences in Effectiveness of CBT on IBS Project 3
Acronym: U54_P3_CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Emeran Mayer, MD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB#20-001118; 1U54DK123755 (NIH)
Record Dates: First submitted 2021-06-11; First posted 2021-12-13 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: IBS - Irritable Bowel Syndrome
Keywords: CBT; MRI; IBS
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: CBT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Treatment Arm (Experimental): Subjects in the "Cognitive Behavioral Treatment" Arm will undergo 8-10 weeks of remote cognitive behavioral therapy. Subjects will complete modules on their phones and will be monitored by study coordinators for support and treatment completion.
  Interventions: Behavioral: COGNITIVE BEHAVIORAL THERAPY
- Usual Care Arm (No Intervention): Subjects in the "Usual Care" Arm will undergo 8-10 weeks of continued lifestyle. Subjects will be asked to report any new medications or lifestyle changes to study coordinators throughout the 8-10 weeks.

INTERVENTIONS:
Behavioral: COGNITIVE BEHAVIORAL THERAPY — 8-10 week self directed on line CBT program approved by FDA
  Arms: Cognitive Behavioral Treatment Arm

SUMMARY:
Cognitive Behavioral Therapy (CBT) is the most well researched and most effective treatment for IBS targeting the brain-gut-microbiome (BGM) axis, and preliminary data show that this therapeutic effect is associated with a reduction of brainstem connectivity with other brain networks.

The increased prevalence of IBS in women, the higher rate of comorbid non-GI pain conditions, as well as the higher prevalence in female IBS of increased sensitivity to a variety of internal and external stimuli (multisensory sensitivity) suggest the presence of important sex differences in some of these BGM mechanisms.

Research performed by UCLA SCOR during previous funding has established an increased responsiveness of the CRF-Locus Coeruleus (LCC) system in female IBS subjects, suggesting that this central noradrenergic brainstem system plays an important role in IBS pathophysiology.

In addition, the study team's earlier research has begun to identify clinical, functional and structural brain mechanisms that may underlie these sex effects. Based on the preliminary data, the overall goal of this project is to use CBT as a probe to study the relationship between specific disease-related alterations of the brain, the gut microbiome, and symptomatic outcome, and identify the role of sex differences in these relationships. Investigators will study male and female IBS patients before and after CBT using the advanced neuroimaging and microbiome technologies of the overall SCOR.

DETAILED DESCRIPTION:
A total of 150 adult IBS participants will be completed in years 1-4 of the proposed studies. These will be 50 males, 50 premenopausal females in the treatment arm (Cognitive behavioral therapy: CBT) and 50 in 'usual care' arm, all bowel habit subtypes.

Screening V1: All subjects will have a pre-screening using a study specific IRB approved prescreening tool (15-20 minutes). lf eligible and interested, the study team will send the ICF via email to the subject and then study team will review the ICF with the subject to determine understanding of study participation and risks/benefits. Subjects will sign and return to the coordinator by electronic/scan/fax methods. The study team will then send participants a short link of preliminary questionnaires via survey Monkey to further determine eligibility for participation and assist the clinician in obtaining accurate medical history as well as assess any risk factors of participation. When determined to be eligible, the study team will set up a video/zoom /phone meeting to complete the initial screening visit/medical and psychological history taking. This will take about 1.5 hour.

Subjects will come to the OCNSR center to complete the study screening, including a physical exam by the RN and RN/NP or MD. Upon arrival, they will date and sign the informed consent and have time to ask any questions. The physical exam will include vital signs, height, weight, and a ROS (review of systems). There will be a single blood sample taken of about 2 teaspoons to determine menstrual cycle (females) and if needed, there may be additional blood (about 1 tablespoon) for IBS-diarrhea or mixed predominance to rule out any other gastrointestinal disease similar to IBS symptoms. Subjects will be given sample collection items to take home for stool and diet diary collection. The stool sample will be collected when they return for the scheduled MRI within 1-3 weeks of screening. They will be given two unique de-identified online Survey Monkey links to complete before the MRI visit. One link is a Diet History Questionnaires (VioScreen) and the other is a group of questionnaires asking about symptoms (IBS), mood and general health and wellbeing. This visit will take about 1.5-2 hours.

MRI V2: Brain and Brainstem Data Acquisition: All participants will undergo a 70 minute structural, resting state, DTI and brain stem MRI scanning session. All subjects will be imaged on a Siemens 3 Tesla Prisma scanner housed at the UCLA Ahmanson-Lovelace Brain Mapping Center (ALBMC). Subjects will complete several state anxiety and symptom-measuring questionnaires upon arrival . Females will need to do daily urine test at home to identify their menstrual phase. When arriving to MRI they will give a urine sample for pregnancy testing and will be excluded if pregnant. A single blood sample will be collected via venipuncture for hormones, cell methylation and pro inflammatory cytokines (15-20 ccs). Subjects will return with their diet diary, stool and saliva (female) sample collections and have all samples reviewed by study coordinator, for viability and collection accuracy.

Scanning will follow parameters of the HBC (Human Brain Connectome) project with anterior and posterior views for each scan. They will have the structural MP Rage (gray matter imaging) scan (time ~14.5 minutes) and subjects can watch a movie of their choice during this scan.

Following this is 2 RSN (resting state) functional scan (total time ~12 minutes). Instructions verbatim are given to subject during the RSN to rest, relax and focus on the crosshair displayed on mirrored screen reflected on the head coil without going to sleep. Following the resting state scan the subject will be asked if they had any pain or discomfort anywhere that may have distracted the subject during the functional resting state and this will be documented on a subject chart.

The next scan is the DTI (diffusion tensor imaging) lasting approximately 10 minutes. Subjects can watch a movie of their choice during this scan.

This visit will take no more than 1.5-2 hours.

Subjects will then be randomized to CBT (66.5 % chance) or usual care (33.5 % chance). The CBT is described below. If usual care, the subject will not have any restrictions on subjects except that the study team will ask subjects not to start new therapies for IBS or new medicines unless it is deemed necessary by their PCP.

CBT: This structured educational and skills based intervention is carried out via internet instruction and individual practice. Subjects will be asked to log into the CBT site once per week for 8-10 weeks with each session lasting between 20 and 40 minutes. The content has been validated in a randomized internet-based CBT trial for IBS. The intervention does not entail any direct therapist contact or interaction with other patients or study participants. The intervention is hosted by Mahana Therapeutics Inc. (named Parallel TM) who is contracted by UCLA to provide the intervention. Following enrollment, each subject will receive a secure login for accessing the CBT site and no personally identifying information will be asked for or passed along to the site or Mahana Therapeutics. During the 8 week intervention period subjects will be contacted by a study coordinator for follow-up should they stop logging in to the web site and they will be able to contact a study coordinator with questions regarding the intervention, website access, etc.

A responder will be defined as a subject with IBS-SSS score change of ≥50 from baseline to end of treatment and corresponds to a clinically meaningful change in symptoms. Participants assigned to the Usual Care condition will have the same questionnaire, neuroimaging, biological and symptom assessments as those in CBT but will not have any specific intervention from the project.

There will be a short mid study SM questionnaire link to complete related to symptoms. After 8-10 weeks of CBT (within 2-3 weeks of completion) they will return for a post-CBT MRI visit identical to description above.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 55 years of age, inclusive.
2. Diagnosis or symptoms of Irritable Bowel Syndrome (IBS) meeting ROME IV diagnostic criteria for IBS (all sub-types).
3. Must be absent of red flags including unexplained weight loss, fevers, anemia or blood in stools.
4. Females must be premenopausal menstruating females. If female and of childbearing potential must be not pregnant, post-partum or breast feeding for at least 6 months. Must have a negative urine test for pregnancy. Must be willing to avoid pregnancy and practice a non-hormonal birth control method such as abstinence, non-hormonal IUD's, or barrier method with spermicide, during the time of study enrollment. Subjects who are on hormonal based birth control (e.g OCP's or implants) will be allowed in the study as long as they still get a monthly menses so menstrual phase can be identified using ovulation kits.
5. Ambulatory outpatient (not depending exclusively on a wheelchair for mobility)
6. Ability to speak the English language fluently due to the standardized assessments involved.

Exclusion Criteria:

1. Evidence of structural abnormality of the gastrointestinal tract. Exclusionary GI conditions include but are not limited to gastrointestinal surgery (exceptions: appendectomy, benign polypectomy, cholecystectomy).
2. Presence of a significant and ongoing medical problem that would interfere with participation in the study or testing the study hypotheses (e.g., major heart disease, neurological disorders, inflammatory diseases such as IBD; esophagitis, celiac disease, gastrointestinal malignancy or obstruction, peptic, duodenal or gastric ulcer disease, etc.). Malignancy (other than localized skin cancer that has been resected) within the previous 5 years.
3. Presence of a major psychiatric diagnosis such as schizophrenia, Bipolar disorder, current ADD diagnosis, Post-traumatic Stress Disorder, Obsessive Compulsive disorder or current history of tobacco or alcohol abuse. Subjects with a history of DSMIV diagnosis of Anxiety or Depression in whom symptoms are not active, will be allowed but noted for post-hoc analysis.
4. Use of investigational drugs, products or devices within 28 days prior to screen and through study participation.
5. Subjects with current regular use of narcotics and or opioids. Use of centrally acting medications that will interfere with the neuroimaging testing (such as systemic steroids, opiate analgesics). Medications which alter GI motility and gastric pH will need to be stopped at least 72 hours prior to any physiologic test visit and during the baseline and treatment intervention. For this we will ask the subject to get approval from their own PCP to stop prior to any intervention. However, rescue medication of bisacodyl and loperamide will be allowed for prolonged constipation and diarrhea, respectively, during intervention periods but not during baseline or within 3 days of follow up MRI. For rescue medication, such as laxatives or antidiarrheal, we will ask to hold off use up to 3 days prior to collecting stool sample.
6. Obesity (BMI >35)
7. Subjects with claustrophobia, metal implants, dental braces, large tattoos (e.g. full arm or back); making MRI safety not possible.
8. History of heavy use of tobacco products or current use of more than 1/3 ppd.
9. Plans to undergo a major medical intervention such a surgery within 6 months of enrollment or during the study, or had major surgery in last 6 months.
10. Current or past history of chronic pain syndrome other than IBS in the IBS group (pain >6 months at any location).
11. Use of antibiotics or probiotics within 3 months of the study enrollment or regular use of probiotics within 4 weeks of enrollment. (enrollment may be deferred)
12. Subjects who currently actively practice CBT or have completed a CBT therapy within 2 years prior to enrolling.
13. Must must have a score of ≥175 (at least moderate severity IBS) on the IB-SSS symptom severity scale completed at screening.
14. Have an average abdominal pain of at least 3 on a 0-10 point scale where 0=no pain and 10=worst imaginable pain.
15. Any other condition that the investigator believes would jeopardize the safety or rights of the subject or would render the subject unable to comply with the study protocol or make use of acquired data non-analyzable.

    -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2021-12-18 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Degree of connectivity between brainstem nuclei and the salience, emotional arousal and sensorimotor networks brain networks. | Through study completion, an average of 5 years
  Degree of connectivity between pre-drawn areas of the brainstem containing pontine nuclei and regions of the salience, emotional arousal, and sensorimotor brain networks will be quantified during a resting state functional MRI scan. The number of significant connections will be determined for pre and post treatment scans for the CBT and usual care conditions and the changes in connectivity following treatment compared for the two conditions.

SECONDARY OUTCOMES:
Abundance of Clostridiales taxa | Through study completion, an average of 5 years
  Stool sample taken pre and post treatment will be processed according to standard laboratory procedures and levels of Clostridiales determined.
Level of tryptophan metabolites | Through study completion, an average of 5 years
  Plasma sample taken pre and post treatment will be processed according to standard laboratory procedures and levels of tryptophan metabolites determined.
KYN/TR ratio. | Through study completion, an average of 5 years
  Plasma samples taken pre and post treatment will be processed according to standard laboratory procedures and KYN/TR ration determined.
Irritable Bowel Symptom Severity scale (IBSSS) | Through study completion, an average of 5 years
  The IBSSS is a validated composite symptom measure for severity of IBS symptoms. It will be used to determine treatment responder (>50 point change pre to post treatment).

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No